CLINICAL TRIAL: NCT02923245
Title: Point-of-Care-Ultrasound Assessment of Bladder Fullness for Girls Awaiting Radiology-Performed Transabdominal Pelvic Ultrasound: A Randomized Controlled Trial
Brief Title: POCUS Assessment of Bladder Fullness for Girls Awaiting Radiology-Performed Transabdominal Pelvic Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Almaz Dessie, Fellow, Pediatric Emergency Medicine, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 744799-9
Record Dates: First submitted 2016-09-24; First posted 2016-10-04 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Abdominal Pain; Pelvic Pain
MeSH Terms: conditions — Abdominal Pain; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- POCUS (Experimental): Patients will be given consecutive IV fluid boluses until a full bladder is visualized by the ED physician on POCUS or the patient endorses maximal bladder fullness on a 0-4 Likert Scale. The patient will then have a transabdominal pelvic ultrasound performed by a radiologist or ultrasound technician.
  Interventions: Other: point-of-care ultrasound
- Usual Care (No Intervention): Patients will be given consecutive IV fluid boluses until the patient endorses sensation of maximum bladder fullness on a 0-4 Likert Scale. The patient will then have a transabdominal pelvic ultrasound performed by a radiologist or ultrasound technician

INTERVENTIONS:
Other: point-of-care ultrasound
  Arms: POCUS

SUMMARY:
The purpose of this study is to assess the accuracy and utility of point-of-care ultrasound (POCUS) of the bladder compared to patient's sensation of bladder fullness in predicting the ability to successfully perform a comprehensive transabdominal pelvic ultrasound in the pediatric Emergency Department (ED). We hypothesize that POCUS can more accurately and more quickly determine adequate bladder fullness to successfully perform transabdominal pelvic ultrasound than patient's perception of bladder fullness.

DETAILED DESCRIPTION:
Ultrasound (US) is the preferred imaging modality in the pediatric ED in the diagnostic evaluation of girls with suspected pelvic pathology. In the transabdominal approach, urine acts as a sonographic acoustic window to image the adnexa and uterus, but this requires a full bladder. Many high acuity pelvic pathologies presenting to the pediatric ED have significant morbidity and mortality associated with delays in diagnosis. Despite this, diagnostic pelvic US is often delayed by the need to fill the bladder, awaiting a patient's report of subjective sensation of bladder fullness. Images of the bladder using POCUS can be easily obtained at the bedside by emergency physicians, providing a quick assessment of the size and shape of the bladder that may be a more accurate, objective measure of bladder fullness. We aim to assess the utility of POCUS of the bladder compared to patient's sensation of bladder fullness in this clinical scenario.

This is a pragmatic, randomized controlled trial of a convenience sample of girls being treated in a pediatric ED who present with an indication for transabdominal pelvic US. Patients will be randomized to two groups:

1. Standard of care group - Patients will be given consecutive IV fluid boluses until sensation of maximum bladder fullness followed by transabdominal pelvic US performed by a radiologist or US technician.
2. Experimental group - Patients will be given consecutive IV fluid boluses until a full bladder is visualized by the ED physician on POCUS followed by transabdominal pelvic US performed by a radiologist or US technician.

Patients in both groups will be assessed at 30-minute intervals for sensation of bladder fullness on a 0-4 Likert Scale, total volume of IVF given per kilogram, and POCUS of the bladder. Overall time between initial ordering of transabdominal pelvic US (Time 0) to the time the patient went for successful US will be recorded and compared between the two groups. Success rate of first attempt at transabdominal pelvic US will also be recorded and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Girls age 8-18 presenting to the pediatric Emergency Department who need transabdominal pelvic ultrasound as determined by their treating providers

Exclusion Criteria:

* History of genitourinary or pelvic anomalies (e.g. neurogenic bladder, urogenital malformation, ambiguous genitalia, Turner Syndrome, ureterocele, bladder diverticulum, imperforate hymen); history of pelvic surgery
* Critically ill patients who are unable to consent
* Sensation of maximal bladder fullness/need to void at time of start of the study
* Nonverbal patients or severe cognitive or language delay

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11-05 (Actual); Study Completion 2016-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hasbro Children's Hospital Emergency Department, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dessie A, Steele D, Liu AR, Amanullah S, Constantine E. Point-of-Care Ultrasound Assessment of Bladder Fullness for Female Patients Awaiting Radiology-Performed Transabdominal Pelvic Ultrasound in a Pediatric Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2018 Nov;72(5):571-580. doi: 10.1016/j.annemergmed.2018.04.010. Epub 2018 Jul 3. PMID 29980460

RESULTS

PARTICIPANT FLOW:
Groups:
- Point-of-care Ultrasound (POCUS): Patients will be given consecutive intravenous (IV) fluid boluses and assessed at 30 minute intervals for sensation of bladder fullness on a 0-4 Likert scale and POCUS assessments of the bladder. Protocol continues until a full bladder is visualized by the emergency department (ED) physician on POCUS or the patient endorses maximal bladder fullness on a 0-4 Likert Scale. The patient will then have a transabdominal pelvic ultrasound performed by a radiologist or ultrasound technician.
  point-of-care ultrasound
- Usual Care (UC): Patients will be given consecutive intravenous (IV) fluid boluses and assessed at 30 minute intervals for sensation of bladder fullness on a 0-4 Likert scale and POCUS assessments of the bladder. Protocol continues until the patient endorses sensation of maximum bladder fullness on a 0-4 Likert Scale. The patient will then have a transabdominal pelvic ultrasound performed by a radiologist or ultrasound technician.
Period: Overall Study
Arm/Group | Point-of-care Ultrasound (POCUS) | Usual Care (UC)
Started | 60 | 60
Completed | 58 | 59
Not Completed | 2 | 1
Not completed — ultrasound order was cancelled | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- POCUS: Patients will be given consecutive IV fluid boluses and assessed at 30 minute intervals for sensation of bladder fullness on a 0-4 Likert scale and POCUS assessments of the bladder. Protocol continues until a full bladder is visualized by the ED physician on POCUS or the patient endorses maximal bladder fullness on a 0-4 Likert Scale. The patient will then have a transabdominal pelvic ultrasound performed by a radiologist or ultrasound technician.
  point-of-care ultrasound
- Usual Care: Patients will be given consecutive IV fluid boluses and assessed at 30 minute intervals for sensation of bladder fullness on a 0-4 Likert scale and POCUS assessments of the bladder. Protocol continues until the patient endorses sensation of maximum bladder fullness on a 0-4 Likert Scale. The patient will then have a transabdominal pelvic ultrasound performed by a radiologist or ultrasound technician.
- Total: Total of all reporting groups
Arm/Group | POCUS | Usual Care | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.43) | 14.7 (2.34) | 14.4 (2.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 31 | 37 | 68
  Non-Hispanic Black | 5 | 5 | 10
  Hispanic | 22 | 14 | 36
  Other | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 120
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 23.0 (4.81) | 25.4 (6.57) | 24.2 (5.86)
Time since last void [Median (Inter-Quartile Range); unit: minutes] | 126.5 [65 to 189] | 120.5 [65 to 200] | 125 [65 to 190]
Time from TAPUS order by physician to study enrollment [Median (Inter-Quartile Range); unit: minutes] | 32.0 [21 to 49.5] | 34.5 [23.5 to 51] | 32.5 [21 to 49.3]
Chief Complaint [Count of Participants; unit: Participants]
  Abdominal Pain | 56 | 50 | 106
  Vomiting | 3 | 3 | 6
  Dysuria/flank pain/hematuria | 5 | 5 | 10
  Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Median Fill-To-Done (FTD) Time
Description: Median time from enrollment to successful completion of TAPUS
Time Frame: on same day as study enrollment
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | POCUS | Usual Care
Number analyzed (Participants) | 58 | 59
minutes | 87.5 [67 to 126] | 139 [92 to 193]
Statistical Analysis 1: Comparison: POCUS vs Usual Care; Test type: Other; Mean Difference (Final Values) = 49.7, 95% CI 2-sided [23.4 to 77.2] — These confidence intervals correspond to the bootstrap analysis

2. Secondary Outcome: Number of Participants Who Had a Successful Transabdominal Pelvic Ultrasound (TAPUS) on First Attempt
Time Frame: on same day as study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POCUS | Usual Care
Number analyzed (Participants) | 58 | 59
Participants | 58 | 50
Statistical Analysis 1: Comparison: POCUS vs Usual Care; Test type: Other; p = 0.006, Test of proportions; Difference in percentages = 15.3, 95% CI 2-sided [5.3 to 25.0]

3. Other Pre Specified Outcome: Number of Participants Receiving IV Narcotics in the Emergency Department
Time Frame: day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POCUS | Usual Care
Number analyzed (Participants) | 58 | 59
Participants | 21 | 26

4. Other Pre Specified Outcome: Total IV Fluids Given Prior to TAPUS
Time Frame: day of enrollment
Measure: Mean (Standard Deviation); unit: ml/Kg
Arm/Group | POCUS | Usual Care
Number analyzed (Participants) | 58 | 59
ml/Kg | 19.4 (15.1) | 22.9 (13.5)

5. Other Pre Specified Outcome: TAPUS Result
Time Frame: day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POCUS | Usual Care
Number analyzed (Participants) | 58 | 59
Participants
  Normal | 46 | 48
  Abnormal | 12 | 11
  Ovarian torsion | 4 | 2
  Simple ovarian cyst | 1 | 3
  Ruptured/hemorrhagic cyst | 5 | 5
  Other ovarian abnormality | 2 | 0
  Uterine anomaly | 0 | 1
  Pathologic free fluid | 1 | 2
  Hydrosalpinx | 1 | 0

6. Other Pre Specified Outcome: Disposition From ED
Time Frame: day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POCUS | Usual Care
Number analyzed (Participants) | 58 | 59
Participants
  Discharged home | 43 | 44
  Admit to ward | 11 | 11
  Admitted to operating room | 5 | 5
  Transferred | 1 | 0

7. Other Pre Specified Outcome: Inter-rater Agreement
Description: Agreement between the POCUS sonographer and the blinded reviewer
Time Frame: at close of study
Population: 304 images were available for assessment of inter-rater reliability
Measure: Number (95% Confidence Interval); unit: weighted kappa
Groups:
- Bladder POCUS Images: all saved POCUS images were de-identified and retrospectively reviewed by the study site's Director of Pediatric Emergency Ultrasound. The reviewer, blinded to the original assessment of the study sonographer, rated each image as small, medium, large, or unidentifiable.
Arm/Group | Bladder POCUS Images
Number analyzed (Participants) | 304
weighted kappa | 0.83 [0.79 to 0.87]

ADVERSE EVENTS:
Arm/Group | POCUS | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes